CLINICAL TRIAL: NCT01662063
Title: A Multicenter Open-Label, Long-Term Extension Study of WA22762 and NA25220 to Evaluate Safety and Efficacy of Subcutaneous Tocilizumab in Patients With Moderate to Severe Rheumatoid Arthritis
Brief Title: A Long-Term Extension Study of WA22762 and NA25220 of Subcutaneous (SC) Tocilizumab (TCZ) in Moderate to Severe Rheumatoid Arthritis (RA)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ML28338
Record Dates: First submitted 2012-07-30; First posted 2012-08-10 (Estimated); Results first posted 2016-10-12 (Estimated); Last update posted 2016-10-12 (Estimated); Status verified 2016-08

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — tocilizumab

ARMS (2):
- SC TCZ QW (Experimental): Participants who received IV TCZ in the previous trial will be switched to SC TCZ 162 mg QW, and those who received SC TCZ will continue at their same dosage of SC TCZ 162 mg QW. Tocilizumab will be given for an additional 96 weeks in this open-label extension study.
  Interventions: Drug: Tocilizumab
- SC TCZ Q2W (Experimental): Participants who received SC TCZ will continue at their same dosage of SC TCZ 162 mg Q2W. Tocilizumab will be given for an additional 96 weeks in this open-label extension study.
  Interventions: Drug: Tocilizumab

INTERVENTIONS:
Drug: Tocilizumab — TCZ will be given as 162 mg SC QW or Q2W for up to 96 weeks.
  Other Names: RoActemra/Actemra

SUMMARY:
This open-label extension study will evaluate the long-term safety and efficacy of SC TCZ in participants with moderate to severe RA who have completed the 97-week WA22762 (NCT01194414) or 96-week NA25220 (NCT01232569) core studies on SC or intravenous (IV) TCZ. Participants will receive TCZ 162 milligrams (mg) SC every week (QW) or every 2 weeks (Q2W) for up to 96 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Completed the 97-week WA22762 (NCT01194414) or 96-week NA25220 (NCT01232569) core study on SC or IV TCZ and, based on the Investigator's judgment, may continue to benefit from TCZ treatment in this study investigating the SC formulation
* Receiving treatment on an outpatient basis
* Females of childbearing potential and males with female partners of childbearing potential must agree to use reliable means of contraception as defined by protocol

Exclusion Criteria:

* Premature withdrawal from WA22762 (NCT01194414) or NA25220 (NCT01232569) core studies for any reason
* History of severe allergic or anaphylactic reactions to human, humanized, or murine monoclonal antibodies
* Evidence of serious uncontrolled concomitant disease or disorder
* Known active current or history of recurrent bacterial, viral, fungal, mycobacterial, or other infections
* Any major episode of infection requiring hospitalization or treatment with IV antibiotics within 4 weeks of Screening or oral antibiotics within 2 weeks of Screening
* History of or currently active primary or secondary immunodeficiency
* Oral corticosteroids at greater than (>) 10 mg per day prednisone or equivalent, or non-steroidal anti-inflammatory drugs (NSAIDs) above the maximum recommended dose
* Intra-articular or parenteral corticosteroids within 4 weeks prior to Baseline
* Treatment with any investigational or commercially available biologic disease-modifying anti-rheumatic drug (DMARD) other than TCZ at any time between completion of the core study WA22762 (NCT01194414) or NA25220 (NCT01232569) and enrollment in the long-term extension study
* Pregnant or breastfeeding women
* History of alcohol, drug, or chemical abuse within 1 year prior to Screening

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 218 (Actual)
Dates: Start 2012-08; Primary Completion 2014-04 (Actual); Study Completion 2014-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Genentech, Inc.
Locations (72):
- United States (71):
  - Tuscaloosa, Alabama
  - Peoria, Arizona
  - Scottsdale, Arizona
  - Tucson, Arizona
  - Fullerton, California
  - Long Beach, California
  - Los Angeles, California
  - San Diego, California
  - San Leandro, California
  - Upland, California
  - Van Nuys, California
  - West Hills, California
  - Whittier, California
  - Denver, Colorado
  - Bridgeport, Connecticut
  - Trumbull, Connecticut
  - Jupiter, Florida
  - Orlando, Florida
  - Palm Harbor, Florida
  - South Miami, Florida
  - Tampa, Florida
  - Venice, Florida
  - Gainesville, Georgia
  - Coeur d'Alene, Idaho
  - Idaho Falls, Idaho
  - Meridian, Idaho
  - Morton Grove, Illinois
  - Springfield, Illinois
  - Vernon Hills, Illinois
  - Wichita, Kansas
  - Monroe, Louisiana
  - Hagerstown, Maryland
  - Wheaton, Maryland
  - Worcester, Massachusetts
  - Saint Claire Shores, Michigan
  - Eagan, Minnesota
  - Flowood, Mississippi
  - Jackson, Mississippi
  - Florissant, Missouri
  - St Louis, Missouri
  - Lincoln, Nebraska
  - Lebanon, New Hampshire
  - Clifton, New Jersey
  - Freehold, New Jersey
  - Manalapan, New Jersey
  - Voorhees Township, New Jersey
  - Albuquerque, New Mexico
  - Albany, New York
  - Brooklyn, New York
  - Orchard Park, New York
  - Asheville, North Carolina
  - Charlotte, North Carolina
  - Raleigh, North Carolina
  - Wilmington, North Carolina
  - Cincinnati, Ohio
  - Perrysburg, Ohio
  - Toledo, Ohio
  - Oklahoma City, Oklahoma
  - Tulsa, Oklahoma
  - Bethlehem, Pennsylvania
  - Duncansville, Pennsylvania
  - Wyomissing, Pennsylvania
  - Charleston, South Carolina
  - Knoxville, Tennessee
  - Memphis, Tennessee
  - Houston, Texas
  - Nassau Bay, Texas
  - Olympia, Washington
  - Seattle, Washington
  - Spokane, Washington
  - Wenatchee, Washington
- Ponce, Puerto Rico

REFERENCES:
- [Derived] Kivitz A, Wallace T, Olech E, Borofsky M, Devenport J, Pei J, Michalska M. Long-Term Safety and Efficacy of Subcutaneously Administered Tocilizumab for Adult Rheumatoid Arthritis: A Multicenter Phase 3b Long-term Extension Study. Rheumatol Ther. 2016 Dec;3(2):291-304. doi: 10.1007/s40744-016-0043-1. Epub 2016 Sep 24. PMID 27747585

RESULTS

PARTICIPANT FLOW:
Groups:
- Subcutaneous (SC) Tocilizumab (TCZ) Every 2 Weeks (Q2W): Participants with moderate to severe rheumatoid arthritis (RA) who completed treatment with SC or intravenous (IV) TCZ in one of the core studies WA22762 (NCT01194414) or NA25220 (NCT01232569) received treatment in this long-term extension (LTE) study for an additional 96 weeks. Participants who received SC TCZ continued at their same dosage of SC TCZ 162 milligrams (mg) Q2W.
- SC TCZ Every Week (QW): Participants with moderate to severe RA who completed treatment with SC or IV TCZ in one of the core studies WA22762 (NCT01194414) or NA25220 (NCT01232569) received treatment in this LTE study for an additional 96 weeks. Participants who received IV TCZ in the previous trial were switched to SC TCZ 162 mg QW, and those who received SC TCZ continued at their same dosage of SC TCZ 162 mg QW.
- Not Treated: Participants with moderate to severe RA who completed treatment with SC or IV TCZ in one of the core studies WA22762 (NCT01194414) or NA25220 (NCT01232569) were enrolled in this LTE study for an additional 96 weeks. Participants who met Screening criteria but did not receive treatment were excluded from analysis and reported in a separate arm.
Period: Overall Study
Arm/Group | Subcutaneous (SC) Tocilizumab (TCZ) Every 2 Weeks (Q2W) | SC TCZ Every Week (QW) | Not Treated
Started | 44 | 173 | 1
Completed | 39 | 144 | 0
Not Completed | 5 | 29 | 1
Not completed — Adverse Event or Intercurrent Illness | 1 | 12 | 0
Not completed — Lack of Efficacy | 1 | 6 | 0
Not completed — Lost to Follow-up | 0 | 4 | 0
Not completed — Protocol Violation | 1 | 0 | 0
Not completed — Withdrawal by Subject | 2 | 4 | 1
Not completed — Physician Decision | 0 | 2 | 0
Not completed — Other | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Safety Population: All participants who received at least one dose of study medication and had at least one post-dose safety assessment.
Groups:
- SC TCZ Q2W: Participants with moderate to severe RA who completed treatment with SC or IV TCZ in one of the core studies WA22762 (NCT01194414) or NA25220 (NCT01232569) received treatment in this LTE study for an additional 96 weeks. Participants who received SC TCZ continued at their same dosage of SC TCZ 162 mg Q2W.
- SC TCZ QW: Participants with moderate to severe RA who completed treatment with SC or IV TCZ in one of the core studies WA22762 (NCT01194414) or NA25220 (NCT01232569) received treatment in this LTE study for an additional 96 weeks. Participants who received IV TCZ in the previous trial were switched to SC TCZ 162 mg QW, and those who received SC TCZ continued at their same dosage of SC TCZ 162 mg QW.
- Total: Total of all reporting groups
Arm/Group | SC TCZ Q2W | SC TCZ QW | Total
Number analyzed (Participants) | 44 | 173 | 217
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.7 (10.18) | 58.1 (10.38) | 58.4 (10.33)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 33 | 133 | 166
  Male | 11 | 40 | 51

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With at Least One Serious Adverse Event (SAE)
Description: Adverse events (AEs) were monitored throughout treatment. AEs were defined as any untoward medical occurrence in a participant who received study drug regardless of causality. SAEs were defined as AEs that were fatal or life-threatening, required hospitalization or prolongation of existing hospitalization, resulted in persistent or significant disability/incapacity, manifested as a congenital anomaly/birth defect, were medically significant, or required intervention to prevent any of the aforementioned outcomes. The number of participants with at least one SAE regardless of treatment relationship was reported.
Time Frame: From Baseline to 8 weeks after last dose; assessed continuously during treatment (up to 96 weeks) and up to 8 weeks after last dose (up to 2 years overall)
Population: Safety Population.
Measure: Number; unit: participants
Arm/Group | SC TCZ Q2W | SC TCZ QW
Number analyzed (Participants) | 44 | 173
participants | 4 | 19

2. Primary Outcome: Percentage of Participants With at Least One SAE
Description: AEs were monitored throughout treatment. AEs were defined as any untoward medical occurrence in a participant who received study drug regardless of causality. SAEs were defined as AEs that were fatal or life-threatening, required hospitalization or prolongation of existing hospitalization, resulted in persistent or significant disability/incapacity, manifested as a congenital anomaly/birth defect, were medically significant, or required intervention to prevent any of the aforementioned outcomes. The percentage of participants with at least one SAE regardless of treatment relationship was calculated.
Time Frame: as for outcome 1
Population: Safety Population.
Measure: Number; unit: percentage of participants
Arm/Group | SC TCZ Q2W | SC TCZ QW
Number analyzed (Participants) | 44 | 173
percentage of participants | 9.1 | 11.0

3. Primary Outcome: Percentage of Participants With a Positive Anti-TCZ Antibody Assay at Any Timepoint
Description: Blood samples were collected to test for the presence of antibodies to TCZ. The percentage of participants with a positive anti-TCZ antibody assay was calculated.
Time Frame: From Baseline to 8 weeks after last dose; assessed at Baseline; Weeks 12, 24, 36, 48, 60, 72, 84, 96; and up to 8 weeks after last dose (up to 2 years overall)
Population: Safety Population; only participants with a valid assay at Screening were included.
Measure: Number; unit: percentage of participants
Arm/Group | SC TCZ Q2W | SC TCZ QW
Number analyzed (Participants) | 44 | 166
percentage of participants | 4.5 | 7.8

4. Primary Outcome: Percentage of Participants With a Positive Anti-TCZ Antibody Assay at Baseline
Description: as for outcome 3
Time Frame: Baseline
Population: Safety Population; only participants with a valid assay at Screening were included.
Measure: Number; unit: percentage of participants
Arm/Group | SC TCZ Q2W | SC TCZ QW
Number analyzed (Participants) | 44 | 166
percentage of participants | 2.3 | 4.8

5. Primary Outcome: Percentage of Participants With a Positive Anti-TCZ Antibody Assay Post-Baseline
Description: Blood samples were collected to test for the presence of antibodies to TCZ. The percentage of participants with a positive anti-TCZ antibody assay was calculated. Positive assay results obtained post-Baseline were further investigated via confirmation assay and a neutralization assay.
Time Frame: From Week 12 up to 8 weeks after last dose; assessed at Weeks 12, 24, 36, 48, 60, 72, 84, 96; and up to 8 weeks after last dose (up to 2 years overall)
Population: Safety Population; only participants with a valid assay at Screening were included.
Measure: Number; unit: percentage of participants
Arm/Group | SC TCZ Q2W | SC TCZ QW
Number analyzed (Participants) | 44 | 166
percentage of participants
  Positive Anti-TCZ Assay | 2.3 | 3.0
  Positive Confirmation Assay | 0 | 0.6
  Positive Neutralizing Assay | 0 | 0.6

6. Secondary Outcome: Percentage of Participants Who Correctly Administered All SC TCZ Doses
Description: Compliance was assessed using drug dispensing logs, diary cards kept by the participant, and return records, as reviewed by the Investigator at regular visits. Total compliance up to the end of treatment was defined as the percentage of participants who correctly administered all scheduled doses of SC TCZ. Correct administration was defined as proper injection technique, injection of the correct amount (162 mg), device not left at room temperature for greater than (>) 8 hours, and absence of other medication errors.
Time Frame: From Baseline to last dose; assessed every 4 weeks during treatment (up to 96 weeks overall)
Population: Intent-to-Treat (ITT) Population: All participants who received at least one dose of study medication and had at least one post-dose efficacy assessment.
Measure: Number; unit: percentage of participants
Arm/Group | SC TCZ Q2W | SC TCZ QW
Number analyzed (Participants) | 44 | 173
percentage of participants | 97.7 | 97.7

7. Secondary Outcome: Disease Activity Score Based on 28 Joints (DAS28) Score
Description: The DAS28 was calculated using the Swollen Joint Count (SJC), Tender Joint Count (TJC), erythrocyte sedimentation rate (ESR), and Global Assessment of Disease Activity by the participant according to Visual Analog Scale (VAS) score. For the DAS28 formula, the SJC and TJC values were based upon 28 joints, and VAS was transformed from a 100-millimeter (mm) scale to a 10-point score. The DAS28 was calculated as (0.56 multiplied by [×] square root of TJC) + (0.28 × square root of SJC) + (0.7 × log natural [ln] ESR) + (0.014 × VAS). Scores may range from 0 to 10, where higher scores indicate increased disease activity.
Time Frame: Baseline and Weeks 12, 24, 36, 48, 60, 72, 84
Population: ITT Population. The "Number of Participants Analyzed" reflects the total number of participants who provided data for the outcome measure. The number of participants who provided data for each analysis (n) is shown in the table.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | SC TCZ Q2W | SC TCZ QW
Number analyzed (Participants) | 44 | 173
units on a scale
  Baseline (n=44,172) | 4.55 (1.732) | 4.60 (1.869)
  Week 12 (n=44,172) | 3.17 (1.443) | 3.42 (1.728)
  Week 24 (n=43,168) | 3.08 (1.351) | 3.35 (1.786)
  Week 36 (n=39,159) | 3.07 (1.425) | 3.29 (1.624)
  Week 48 (n=18,141) | 3.15 (1.392) | 3.25 (1.639)
  Week 60 (n=2,92) | 4.10 (0.515) | 3.12 (1.626)
  Week 72 (n=1,52) | 5.76 (NA) — Standard deviation could not be calculated because the analysis only included 1 participant. | 3.05 (1.970)
  Week 84 (n=0,11) | NA (NA) — No participants provided evaluable data for the analysis. | 2.78 (1.434)

8. Secondary Outcome: Change From Baseline in DAS28 Score
Description: The DAS28 was calculated using the SJC, TJC, ESR, and Global Assessment of Disease Activity by the participant according to VAS score. For the DAS28 formula, the SJC and TJC values were based upon 28 joints, and VAS was transformed from a 100-mm scale to a 10-point score. The DAS28 was calculated as (0.56 × square root of TJC) + (0.28 × square root of SJC) + (0.7 × ln ESR) + (0.014 × VAS). Scores may range from 0 to 10, where higher scores indicate increased disease activity. The change from Baseline to each visit was calculated, where positive changes represent an increase or worsening in disease activity.
Time Frame: Baseline to Weeks 12, 24, 36, 48, 60, 72, 84
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | SC TCZ Q2W | SC TCZ QW
Number analyzed (Participants) | 44 | 172
units on a scale
  Week 12 (n=44,171) | -1.38 (1.522) | -1.19 (1.415)
  Week 24 (n=43,167) | -1.42 (1.383) | -1.23 (1.692)
  Week 36 (n=39,158) | -1.51 (1.312) | -1.29 (1.429)
  Week 48 (n=18,140) | -1.66 (1.340) | -1.32 (1.538)
  Week 60 (n=2,91) | 0.65 (1.410) | -1.29 (1.286)
  Week 72 (n=1,52) | -0.35 (NA) — Standard deviation could not be calculated because the analysis only included 1 participant. | -1.53 (1.435)
  Week 84 (n=0,10) | NA (NA) — No participants provided evaluable data for the analysis. | -1.57 (1.312)

9. Secondary Outcome: Clinical Disease Activity Index (CDAI) Score
Description: The CDAI was calculated using the SJC, TJC, and Global Assessment of Disease Activity by the patient and by the physician according to separate VAS scores. For the CDAI formula, the SJC and TJC values were based upon 28 joints, and VAS was transformed from a 100-mm scale to a 10-point score. The CDAI was calculated as the sum of the component scores, that is, SJC + TJC + VAS (participant) + VAS (physician). Scores may range from 0 to 76, where higher scores indicate increased disease activity.
Time Frame: Baseline and Weeks 12, 24, 36, 48, 60, 72, 84
Population: ITT Population; only those participants who provided evaluable data (n) were included in the analysis.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | SC TCZ Q2W | SC TCZ QW
Number analyzed (Participants) | 44 | 173
units on a scale
  Baseline (n=44,173) | 20.10 (15.467) | 23.91 (16.346)
  Week 12 (n=44,172) | 13.99 (13.058) | 18.19 (14.145)
  Week 24 (n=42,166) | 14.86 (13.232) | 18.03 (13.665)
  Week 36 (n=39,159) | 13.26 (11.839) | 16.92 (12.598)
  Week 48 (n=18,140) | 15.81 (16.479) | 16.55 (13.559)
  Week 60 (n=2,92) | 13.60 (2.828) | 14.71 (11.954)
  Week 72 (n=1,52) | 27.80 (NA) — Standard deviation could not be calculated because the analysis only included 1 participant. | 16.04 (15.476)
  Week 84 (n=0,11) | NA (NA) — No participants provided evaluable data for the analysis | 12.82 (9.154)

10. Secondary Outcome: Change From Baseline in CDAI Score
Description: The CDAI was calculated using the SJC, TJC, and Global Assessment of Disease Activity by the patient and by the physician according to separate VAS scores. For the CDAI formula, the SJC and TJC values were based upon 28 joints, and VAS was transformed from a 100-mm scale to a 10-point score. The CDAI was calculated as the sum of the component scores, that is, SJC + TJC + VAS (participant) + VAS (physician). Scores may range from 0 to 76, where higher scores indicate increased disease activity. The change from Baseline to each visit was calculated, where positive changes represent an increase or worsening in disease activity.
Time Frame: Baseline to Weeks 12, 24, 36, 48, 60, 72, 84
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | SC TCZ Q2W | SC TCZ QW
Number analyzed (Participants) | 44 | 173
units on a scale
  Week 12 (n=44,172) | -6.11 (13.219) | -5.81 (12.010)
  Week 24 (n=42,166) | -5.23 (14.134) | -5.47 (13.754)
  Week 36 (n=39,159) | -7.00 (12.266) | -6.63 (10.676)
  Week 48 (n=18,140) | -6.63 (13.479) | -6.70 (12.328)
  Week 60 (n=2,92) | -14.05 (20.294) | -7.05 (11.065)
  Week 72 (n=1,52) | -16.20 (NA) — Standard deviation could not be calculated because the analysis only included 1 participant. | -6.31 (12.999)
  Week 84 (n=0,11) | NA (NA) — No participants provided evaluable data for the analysis | -10.01 (18.580)

11. Secondary Outcome: Simplified Disease Activity Index (SDAI) Score
Description: The SDAI was calculated using the SJC, TJC, Global Assessment of Disease Activity by the patient and by the physician according to separate VAS scores, and high-sensitivity C-reactive protein (hsCRP) level. For the SDAI formula, the SJC and TJC values were based upon 28 joints, and VAS was transformed from a 100-mm scale to a 10-point score. The SDAI was calculated as the sum of the component scores, that is, SJC + TJC + VAS (participant) + VAS (physician) + hsCRP. Because the formula includes hsCRP, scores may theoretically range from 0 to infinity, where higher scores indicate increased disease activity. However, based upon normal hsCRP level within 1 milligram per deciliter (mg/dL), scores would be expected to fall within less than or equal to (≤) 77 points.
Time Frame: Baseline and Weeks 12, 24, 36, 48, 60, 72, 84
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | SC TCZ Q2W | SC TCZ QW
Number analyzed (Participants) | 44 | 173
units on a scale
  Baseline (n=44,170) | 21.54 (15.717) | 25.10 (16.972)
  Week 12 (n=44,172) | 14.48 (13.058) | 18.32 (14.199)
  Week 24 (n=41,166) | 15.42 (13.266) | 18.18 (13.779)
  Week 36 (n=39,159) | 13.75 (11.841) | 17.06 (12.621)
  Week 48 (n=18,140) | 15.85 (16.490) | 16.76 (13.603)
  Week 60 (n=2,92) | 13.63 (2.841) | 14.90 (12.045)
  Week 72 (n=1,52) | 27.82 (NA) — Standard deviation could not be calculated because the analysis only included 1 participant. | 16.23 (15.730)
  Week 84 (n=0,11) | NA (NA) — No participants provided evaluable data for the analysis | 12.90 (9.163)

12. Secondary Outcome: Change From Baseline in SDAI Score
Description: The SDAI was calculated using the SJC, TJC, Global Assessment of Disease Activity by the patient and by the physician according to separate VAS scores, and hsCRP level. For the SDAI formula, the SJC and TJC values were based upon 28 joints, and VAS was transformed from a 100-mm scale to a 10-point score. The SDAI was calculated as the sum of the component scores, that is, SJC + TJC + VAS (participant) + VAS (physician) + hsCRP. Because the formula includes hsCRP, scores may theoretically range from 0 to infinity, where higher scores indicate increased disease activity. However, based upon normal hsCRP level within 1 mg/dL, scores would be expected to fall within ≤77 points. The change from Baseline to each visit was calculated, where positive changes represent an increase or worsening in disease activity.
Time Frame: Baseline to Weeks 12, 24, 36, 48, 60, 72, 84
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | SC TCZ Q2W | SC TCZ QW
Number analyzed (Participants) | 44 | 170
units on a scale
  Week 12 (n=44,169) | -7.07 (13.671) | -7.00 (12.056)
  Week 24 (n=41,163) | -5.71 (14.217) | -6.79 (13.069)
  Week 36 (n=39,157) | -7.99 (12.858) | -7.38 (10.953)
  Week 48 (n=18,139) | -8.17 (14.640) | -7.29 (12.454)
  Week 60 (n=2,91) | -14.46 (20.873) | -7.52 (10.846)
  Week 72 (n=1,52) | -17.04 (NA) — Standard deviation could not be calculated because the analysis only included 1 participant. | -7.10 (13.379)
  Week 84 (n=0,10) | NA (NA) — No participants provided evaluable data for the analysis | -9.48 (19.290)

13. Secondary Outcome: Tender Joint Count (TJC) Score
Description: Sixty-eight joints were assessed and classified as tender/not tender by pressure and joint manipulation on physical examination. The number of tender joints was taken as the TJC score, where values may range from 0 to 68.
Time Frame: Baseline and Weeks 12, 24, 36, 48, 60, 72, 84
Population: ITT Population; only those participants who provided evaluable data (n) were included in the analysis.
Measure: Mean (Standard Deviation); unit: tender joints
Arm/Group | SC TCZ Q2W | SC TCZ QW
Number analyzed (Participants) | 44 | 173
tender joints
  Baseline (n=44,173) | 13.84 (13.883) | 19.14 (18.469)
  Week 12 (n=44,172) | 9.86 (11.727) | 14.06 (14.874)
  Week 24 (n=42,167) | 10.95 (14.221) | 13.86 (15.176)
  Week 36 (n=39,159) | 9.10 (11.392) | 13.45 (14.398)
  Week 48 (n=18,141) | 10.61 (14.825) | 12.85 (16.192)
  Week 60 (n=2,92) | 5.50 (0.707) | 10.47 (12.589)
  Week 72 (n=1,52) | 21.00 (NA) — Standard deviation could not be calculated because the analysis only included 1 participant. | 11.38 (15.444)
  Week 84 (n=0,11) | NA (NA) — No participants provided evaluable data for the analysis | 9.36 (10.984)

14. Secondary Outcome: Change From Baseline in TJC Score
Description: Sixty-eight joints were assessed and classified as tender/not tender by pressure and joint manipulation on physical examination. The number of tender joints was taken as the TJC score, where values may range from 0 to 68. The change from Baseline to each visit was calculated, where positive changes represent an increase in number of tender joints.
Time Frame: Baseline to Weeks 12, 24, 36, 48, 60, 72, 84
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: tender joints
Arm/Group | SC TCZ Q2W | SC TCZ QW
Number analyzed (Participants) | 44 | 173
tender joints
  Week 12 (n=44,172) | -3.98 (12.082) | -5.17 (12.175)
  Week 24 (n=42,167) | -2.69 (12.546) | -5.12 (14.817)
  Week 36 (n=39,159) | -4.03 (10.559) | -5.60 (12.402)
  Week 48 (n=18,141) | -4.00 (12.902) | -5.95 (13.899)
  Week 60 (n=2,92) | -9.00 (12.728) | -6.23 (10.672)
  Week 72 (n=1,52) | -3.00 (NA) — Standard deviation could not be calculated because the analysis only included 1 participant. | -4.98 (11.514)
  Week 84 (n=0,11) | NA (NA) — No participants provided evaluable data for the analysis | -6.27 (13.835)

15. Secondary Outcome: Swollen Joint Count (SJC) Score
Description: Sixty-six joints were assessed and classified as swollen/not swollen by pressure and joint manipulation on physical examination. The number of swollen joints was taken as the SJC score, where values may range from 0 to 66.
Time Frame: Baseline and Weeks 12, 24, 36, 48, 60, 72, 84
Population: ITT Population; only those participants who provided evaluable data (n) were included in the analysis.
Measure: Mean (Standard Deviation); unit: swollen joints
Arm/Group | SC TCZ Q2W | SC TCZ QW
Number analyzed (Participants) | 44 | 173
swollen joints
  Baseline (n=44,173) | 9.07 (8.877) | 10.83 (10.855)
  Week 12 (n=44,172) | 5.61 (7.144) | 7.87 (8.839)
  Week 24 (n=42,167) | 5.98 (8.587) | 8.57 (8.783)
  Week 36 (n=39,159) | 5.51 (8.398) | 6.92 (7.055)
  Week 48 (n=18,141) | 4.78 (9.078) | 7.23 (7.870)
  Week 60 (n=2,92) | 2.00 (2.828) | 6.52 (7.184)
  Week 72 (n=1,52) | 2.00 (NA) — Standard deviation could not be calculated because the analysis only included 1 participant. | 7.98 (8.873)
  Week 84 (n=0,11) | NA (NA) — No participants provided evaluable data for the analysis | 8.64 (8.857)

16. Secondary Outcome: Change From Baseline in SJC Score
Description: Sixty-six joints were assessed and classified as swollen/not swollen by pressure and joint manipulation on physical examination. The number of swollen joints was taken as the SJC score, where values may range from 0 to 66. The change from Baseline to each visit was calculated, where positive changes represent an increase in number of swollen joints.
Time Frame: Baseline to Weeks 12, 24, 36, 48, 60, 72, 84
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: swollen joints
Arm/Group | SC TCZ Q2W | SC TCZ QW
Number analyzed (Participants) | 44 | 173
swollen joints
  Week 12 (n=44,172) | -3.45 (7.026) | -3.00 (8.543)
  Week 24 (n=42,167) | -3.45 (8.434) | -2.31 (9.162)
  Week 36 (n=39,159) | -3.33 (6.868) | -3.89 (8.134)
  Week 48 (n=18,141) | -6.56 (9.332) | -3.25 (9.543)
  Week 60 (n=2,92) | -8.50 (12.021) | -3.20 (8.702)
  Week 72 (n=1,52) | -15.00 (NA) — Standard deviation could not be calculated because the analysis only included 1 participant. | -1.15 (10.114)
  Week 84 (n=0,11) | NA (NA) — No participants provided evaluable data for the analysis | -2.64 (13.493)

17. Secondary Outcome: Number of Participants With a Disease-Modifying Anti-Rheumatic Drug (DMARD) Dose Reduction, Interruption, or Discontinuation
Description: Use of concomitant medications, including non-biologic DMARDs, was recorded throughout the study. Any change in DMARD therapy was documented and reported among those participants receiving at least one DMARD at Baseline.
Time Frame: From Baseline to last dose; assessed every 4 weeks during treatment (up to 96 weeks overall)
Population: ITT Population; only participants receiving at least one DMARD at Baseline were included.
Measure: Number; unit: participants
Arm/Group | SC TCZ Q2W | SC TCZ QW
Number analyzed (Participants) | 41 | 161
participants
  Any Dose Reduction/Interruption/Discontinuation | 3 | 37
  Dose Reduction | 1 | 14
  Dose Interruption ≤60 Days | 1 | 15
  Dose Reduction/Interruption ≤60 Days | 1 | 27
  Discontinuation >60 Days | 2 | 15

18. Secondary Outcome: Percentage of Participants With a DMARD Dose Reduction, Interruption, or Discontinuation
Description: as for outcome 17
Time Frame: From Baseline to last dose; assessed every 4 weeks during treatment (up to 96 weeks overall)
Population: ITT Population; only participants receiving at least one DMARD at Baseline were included.
Measure: Number; unit: percentage of participants
Arm/Group | SC TCZ Q2W | SC TCZ QW
Number analyzed (Participants) | 41 | 161
percentage of participants
  Any Dose Reduction/Interruption/Discontinuation | 7.3 | 23.0
  Dose Reduction | 2.4 | 8.7
  Dose Interruption ≤60 Days | 2.4 | 9.3
  Dose Reduction/Interruption ≤60 Days | 2.4 | 16.8
  Discontinuation >60 Days | 4.9 | 9.3

19. Secondary Outcome: Percentage of Reasons Given for DMARD Dose Reduction or Interruption
Description: Use of concomitant medications, including non-biologic DMARDs, was recorded throughout the study. Any change in DMARD therapy was documented and reported among those participants receiving at least one DMARD at Baseline. The reasons for any DMARD dose reduction/interruption ≤60 days were reported. More than one reason could be given for a single change in DMARD therapy, and each participant could also change DMARD therapy more than once. Therefore, the number of reasons could exceed the number of participants analyzed.
Time Frame: From Baseline to last dose; assessed every 4 weeks during treatment (up to 96 weeks overall)
Population: ITT Population; only participants with a DMARD dose reduction/interruption ≤60 days were included.
Measure: Number; unit: percentage of reasons
Units Other Than Participants: Reasons
Arm/Group | SC TCZ Q2W | SC TCZ QW
Number analyzed (Participants) | 1 | 27
Number analyzed (Reasons) | 2 | 41
percentage of reasons
  AEs | 0 | 70.7
  Efficacy | 0 | 2.4
  Joint Surgery | 0 | 2.4
  Medical History | 100.0 | 2.4
  RA Improvement | 0 | 7.3
  RA Treatment | 0 | 2.4
  Replace Previous Drug | 0 | 2.4
  Participant Request | 0 | 2.4
  Not Specified | 0 | 7.3

20. Secondary Outcome: Percentage of Reasons Given for DMARD Discontinuation
Description: Use of concomitant medications, including non-biologic DMARDs, was recorded throughout the study. Any change in DMARD therapy was documented and reported among those participants receiving at least one DMARD at Baseline. The reasons for any DMARD discontinuation were reported. More than one reason could be given for a single change in DMARD therapy, and each participant could also change DMARD therapy more than once. Therefore, the number of reasons could exceed the number of participants analyzed.
Time Frame: From Baseline to last dose; assessed every 4 weeks during treatment (up to 96 weeks overall)
Population: ITT Population; only participants with a DMARD discontinuation >60 days were included.
Measure: Number; unit: percentage of reasons
Units Other Than Participants: Reasons
Arm/Group | SC TCZ Q2W | SC TCZ QW
Number analyzed (Participants) | 2 | 15
Number analyzed (Reasons) | 3 | 16
percentage of reasons
  AEs | 66.7 | 43.8
  Efficacy | 33.3 | 0
  Investigator Recommendation | 0 | 6.3
  RA Improvement | 0 | 31.3
  Participant Request | 0 | 6.3
  Too Expensive | 0 | 6.3
  Not Specified | 0 | 6.3

21. Secondary Outcome: Number of Participants With a Corticosteroid (CCS) Dose Reduction, Interruption, or Discontinuation
Description: Use of concomitant medications, including CCS treatment, was recorded throughout the study. Any change in CCS therapy was documented and reported among those participants who received at least one CCS before the last dose of SC TCZ.
Time Frame: From Baseline to last dose; assessed every 4 weeks during treatment (up to 96 weeks overall)
Population: ITT Population; only participants who received at least one CCS before the last dose of TCZ were included.
Measure: Number; unit: participants
Arm/Group | SC TCZ Q2W | SC TCZ QW
Number analyzed (Participants) | 15 | 89
participants
  Any Dose Reduction/Interruption/Discontinuation | 6 | 33
  Dose Reduction | 5 | 24
  Dose Interruption ≤14 Days | 0 | 2
  Discontinuation >14 Days | 2 | 19

22. Secondary Outcome: Percentage of Participants With a CCS Dose Reduction, Interruption, or Discontinuation
Description: as for outcome 21
Time Frame: From Baseline to last dose; assessed every 4 weeks during treatment (up to 96 weeks overall)
Population: ITT Population; only participants who received at least one CCS before the last dose of TCZ were included.
Measure: Number; unit: percentage of participants
Arm/Group | SC TCZ Q2W | SC TCZ QW
Number analyzed (Participants) | 15 | 89
percentage of participants
  Any Dose Reduction/Interruption/Discontinuation | 40.0 | 37.1
  Dose Reduction | 33.3 | 27.0
  Dose Interruption ≤14 Days | 0 | 2.2
  Discontinuation >14 Days | 13.3 | 21.3

23. Secondary Outcome: Percentage of Reasons Given for CCS Dose Reduction
Description: Use of concomitant medications, including CCS treatment, was recorded throughout the study. Any change in CCS therapy was documented and reported among those participants who received at least one CCS before the last dose of SC TCZ. The reasons for any CCS dose reduction were reported. More than one reason could be given for a single change in CCS therapy, and each participant could also change CCS therapy more than once. Therefore, the number of reasons could exceed the number of participants analyzed.
Time Frame: From Baseline to last dose; assessed every 4 weeks during treatment (up to 96 weeks overall)
Population: ITT Population; only participants with a CCS dose reduction were included.
Measure: Number; unit: percentage of reasons
Units Other Than Participants: Reasons
Arm/Group | SC TCZ Q2W | SC TCZ QW
Number analyzed (Participants) | 5 | 24
Number analyzed (Reasons) | 14 | 84
percentage of reasons
  AEs | 0 | 3.6
  Medical History | 42.9 | 0
  RA Treatment | 0 | 2.4
  Steroid Tapering | 50.0 | 91.7
  Participant Request | 0 | 1.2
  Not Specified | 7.1 | 1.2

24. Secondary Outcome: Percentage of Reasons Given for CCS Dose Interruption
Description: Use of concomitant medications, including CCS treatment, was recorded throughout the study. Any change in CCS therapy was documented and reported among those participants who received at least one CCS before the last dose of SC TCZ. The reasons for any CCS dose interruption ≤14 days were reported. More than one reason could be given for a single change in CCS therapy, and each participant could also change CCS therapy more than once. Therefore, the number of reasons could exceed the number of participants analyzed.
Time Frame: From Baseline to last dose; assessed every 4 weeks during treatment (up to 96 weeks overall)
Population: ITT Population; only participants with a CCS dose interruption ≤14 days were included. Results were only reported for the QW arm because no participants in the Q2W arm had a CCS dose interruption.
Measure: Number; unit: percentage of reasons
Units Other Than Participants: Reasons
Arm/Group | SC TCZ QW
Number analyzed (Participants) | 2
Number analyzed (Reasons) | 3
percentage of reasons
  Hospitalization | 33.3
  Steroid Tapering | 66.7

25. Secondary Outcome: Percentage of Reasons Given for CCS Discontinuation
Description: Use of concomitant medications, including CCS treatment, was recorded throughout the study. Any change in CCS therapy was documented and reported among those participants who received at least one CCS before the last dose of SC TCZ. The reasons for any CCS discontinuation >14 days were reported. More than one reason could be given for a single change in CCS therapy, and each participant could also change CCS therapy more than once. Therefore, the number of reasons could exceed the number of participants analyzed.
Time Frame: From Baseline to last dose; assessed every 4 weeks during treatment (up to 96 weeks overall)
Population: ITT Population; only participants with a CCS discontinuation >14 days were included.
Measure: Number; unit: percentage of reasons
Units Other Than Participants: Reasons
Arm/Group | SC TCZ Q2W | SC TCZ QW
Number analyzed (Participants) | 2 | 19
Number analyzed (Reasons) | 2 | 27
percentage of reasons
  AE Resolution | 0 | 18.5
  AEs | 50.0 | 11.1
  Prescription End | 0 | 14.8
  RA Improvement | 0 | 14.8
  Steroid Tapering | 50.0 | 18.5
  Participant Request | 0 | 7.4
  Not Specified | 0 | 14.8

26. Secondary Outcome: Number of Participants Who Switched From the QW Regimen and Remained on the Q2W Regimen
Description: Participants could switch between regimens at the Investigator's judgment based upon safety, efficacy, and pharmacokinetic/pharmacodynamic data. The number of participants who switched from the QW to the Q2W regimen and did not return to the QW regimen was reported.
Time Frame: From Baseline to last dose; assessed every 4 weeks during treatment (up to 96 weeks overall)
Population: ITT Population. The results were presented for all participants to account for multiple switches between arms (i.e., participants who started in the Q2W arm could have switched to QW and then switched back to Q2W, making them analyzable for the outcome measure).
Measure: Number; unit: participants
Groups:
- SC TCZ/All Participants: Participants with moderate to severe RA who completed treatment with SC or IV TCZ in one of the core studies WA22762 (NCT01194414) or NA25220 (NCT01232569) received treatment in this LTE study for an additional 96 weeks. Participants who received IV TCZ in the previous trial were switched to SC TCZ 162 mg QW, and those who received SC TCZ continued at their same dosage of SC TCZ 162 mg QW or SC TCZ 162 mg Q2W.
Arm/Group | SC TCZ/All Participants
Number analyzed (Participants) | 217
participants | 14

27. Secondary Outcome: Percentage of Participants Who Switched From the QW Regimen and Remained on the Q2W Regimen
Description: Participants could switch between regimens at the Investigator's judgment based upon safety, efficacy, and pharmacokinetic/pharmacodynamic data. The percentage of participants who switched from the QW to the Q2W regimen and did not return to the QW regimen was calculated.
Time Frame: From Baseline to last dose; assessed every 4 weeks during treatment (up to 96 weeks overall)
Population: as for outcome 26
Measure: Number; unit: percentage of participants
Arm/Group | SC TCZ/All Participants
Number analyzed (Participants) | 217
percentage of participants | 6.5

28. Secondary Outcome: Number of Participants Who Returned to the QW Regimen After Switching to the Q2W Regimen
Description: Participants could switch between regimens at the Investigator's judgment based upon safety, efficacy, and pharmacokinetic/pharmacodynamic data. The number of participants who switched from the QW to the Q2W regimen and thereafter returned to the QW regimen was reported with the reason for returning to the QW regimen.
Time Frame: From Baseline to last dose; assessed every 4 weeks during treatment (up to 96 weeks overall)
Population: ITT Population; only participants who switched from the QW to Q2W regimen were included.
Measure: Number; unit: participants
Arm/Group | SC TCZ/All Participants
Number analyzed (Participants) | 15
participants
  Any Reason | 1
  Investigator Recommendation | 1

29. Secondary Outcome: Time to Return to the QW Regimen After Switching to the Q2W Regimen
Description: Participants could switch between regimens at the Investigator's judgment based upon safety, efficacy, and pharmacokinetic/pharmacodynamic data. Time to return was defined as the time between switching to the Q2W regimen and returning to the previous QW regimen.
Time Frame: From Baseline to last dose; assessed every 4 weeks during treatment (up to 96 weeks overall)
Population: ITT Population; only participants who switched from the QW to Q2W regimen and returned to the QW regimen were included.
Measure: Median (Full Range); unit: weeks
Arm/Group | SC TCZ/All Participants
Number analyzed (Participants) | 1
weeks | 20

30. Secondary Outcome: Global Assessment of Disease Activity by the Participant According to Visual Analog Scale (VAS) Score
Description: The Global Assessment of Disease Activity was performed using a 100-mm horizontal VAS. Scores may range from 0 mm ("no disease activity") to 100 mm ("maximum disease activity"), with higher scores representing an increase in perceived symptoms.
Time Frame: Baseline and Weeks 12, 24, 36, 48, 60, 72, 84
Population: ITT Population; only those participants who provided evaluable data (n) were included in the analysis.
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | SC TCZ Q2W | SC TCZ QW
Number analyzed (Participants) | 44 | 173
mm
  Baseline (n=44,173) | 39.39 (24.483) | 47.25 (29.868)
  Week 12 (n=44,172) | 31.80 (23.878) | 37.84 (28.130)
  Week 24 (n=43,168) | 31.86 (25.639) | 37.51 (27.536)
  Week 36 (n=39,159) | 30.13 (23.345) | 37.44 (27.519)
  Week 48 (n=18,141) | 37.95 (24.878) | 34.63 (27.136)
  Week 60 (n=2,92) | 54.00 (24.042) | 32.86 (27.932)
  Week 72 (n=1,52) | 57.00 (NA) — Standard deviation could not be calculated because the analysis only included 1 participant. | 30.83 (28.425)
  Week 84 (n=0,11) | NA (NA) — No participants provided evaluable data for the analysis | 30.00 (26.348)

31. Secondary Outcome: Change From Baseline in Global Assessment of Disease Activity by the Participant According to VAS Score
Description: The Global Assessment of Disease Activity was performed using a 100-mm horizontal VAS. Scores may range from 0 mm ("no disease activity") to 100 mm ("maximum disease activity"), with higher scores representing an increase in perceived symptoms. The change from Baseline to each visit was calculated, where positive changes represent an increase or worsening in perceived disease activity.
Time Frame: Baseline to Weeks 12, 24, 36, 48, 60, 72, 84
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | SC TCZ Q2W | SC TCZ QW
Number analyzed (Participants) | 44 | 173
mm
  Week 12 (n=44,172) | -7.59 (22.689) | -9.59 (22.348)
  Week 24 (n=43,168) | -6.67 (18.977) | -9.67 (26.260)
  Week 36 (n=39,159) | -11.59 (23.736) | -10.14 (25.338)
  Week 48 (n=18,141) | -5.61 (21.892) | -11.47 (25.839)
  Week 60 (n=2,92) | 11.50 (30.406) | -9.93 (22.992)
  Week 72 (n=1,52) | 19.00 (NA) — Standard deviation could not be calculated because the analysis only included 1 participant. | -13.82 (25.779)
  Week 84 (n=0,11) | NA (NA) — No participants provided evaluable data for the analysis | -10.82 (19.778)

32. Secondary Outcome: Global Assessment of Pain by the Participant According to VAS Score
Description: The Global Assessment of Pain was performed using a 100-mm horizontal VAS. Scores may range from 0 mm ("no pain") to 100 mm ("unbearable pain"), with higher scores representing an increase in pain.
Time Frame: Baseline and Weeks 12, 24, 36, 48, 60, 72, 84
Population: ITT Population; only those participants who provided evaluable data (n) were included in the analysis.
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | SC TCZ Q2W | SC TCZ QW
Number analyzed (Participants) | 44 | 173
mm
  Baseline (n=44,173) | 36.89 (23.044) | 45.42 (29.448)
  Week 12 (n=44,172) | 29.30 (22.782) | 33.27 (25.984)
  Week 24 (n=43,168) | 29.42 (24.509) | 34.48 (24.841)
  Week 36 (n=39,159) | 28.38 (20.607) | 34.40 (25.149)
  Week 48 (n=18,141) | 33.44 (21.742) | 31.52 (25.892)
  Week 60 (n=2,92) | 50.00 (14.142) | 30.94 (27.635)
  Week 72 (n=1,52) | 42.00 (NA) — Standard deviation could not be calculated because the analysis only included 1 participant. | 29.20 (26.733)
  Week 84 (n=0,11) | NA (NA) — No participants provided evaluable data for the analysis | 25.36 (25.598)

33. Secondary Outcome: Change From Baseline in Global Assessment of Pain by the Participant According to VAS Score
Description: The Global Assessment of Pain was performed using a 100-mm horizontal VAS. Scores may range from 0 mm ("no pain") to 100 mm ("unbearable pain"), with higher scores representing an increase in pain. The change from Baseline to each visit was calculated, where positive changes represent an increase or worsening in pain.
Time Frame: Baseline to Weeks 12, 24, 36, 48, 60, 72, 84
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | SC TCZ Q2W | SC TCZ QW
Number analyzed (Participants) | 44 | 173
mm
  Week 12 (n=44,172) | -7.59 (22.145) | -12.27 (21.582)
  Week 24 (n=43,168) | -6.63 (20.641) | -10.76 (24.154)
  Week 36 (n=39,159) | -10.62 (22.783) | -10.91 (22.747)
  Week 48 (n=18,141) | -8.00 (18.166) | -12.91 (24.950)
  Week 60 (n=2,92) | 3.00 (25.456) | -10.07 (22.001)
  Week 72 (n=1,52) | 3.00 (NA) — Standard deviation could not be calculated because the analysis only included 1 participant. | -12.47 (23.522)
  Week 84 (n=0,11) | NA (NA) — No participants provided evaluable data for the analysis | -14.64 (20.911)

34. Secondary Outcome: Heath Assessment Questionnaire-Disability Index (HAQ-DI) Score
Description: The Stanford HAQ-DI was calculated as the average of 20 questions, each scored from 0 (no difficulty) to 3 (unable to do). The questionnaire included 8 component sets: dressing/grooming, arising, eating, walking, hygiene, reach, grip, and common activities. Overall scores may range from 0 to 3, with higher scores representing increased disability.
Time Frame: Baseline and Weeks 12, 24, 36, 48, 60, 72, 84
Population: ITT Population; only those participants who provided evaluable data (n) were included in the analysis.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | SC TCZ Q2W | SC TCZ QW
Number analyzed (Participants) | 44 | 173
units on a scale
  Baseline (n=44,173) | 0.98 (0.682) | 1.20 (0.729)
  Week 12 (n=44,172) | 0.95 (0.688) | 1.11 (0.750)
  Week 24 (n=43,167) | 0.94 (0.717) | 1.09 (0.725)
  Week 36 (n=39,159) | 0.95 (0.682) | 1.10 (0.741)
  Week 48 (n=18,141) | 0.97 (0.596) | 1.04 (0.745)
  Week 60 (n=2,92) | 2.13 (0.530) | 1.01 (0.779)
  Week 72 (n=1,52) | 2.25 (NA) — Standard deviation could not be calculated because the analysis only included 1 participant. | 0.97 (0.844)
  Week 84 (n=0,11) | NA (NA) — No participants provided evaluable data for the analysis. | 1.14 (0.730)

35. Secondary Outcome: Change From Baseline in HAQ-DI Score
Description: The Stanford HAQ-DI was calculated as the average of 20 questions, each scored from 0 (no difficulty) to 3 (unable to do). The questionnaire included 8 component sets: dressing/grooming, arising, eating, walking, hygiene, reach, grip, and common activities. Overall scores may range from 0 to 3, with higher scores representing increased disability. The change from Baseline to each visit was calculated, where positive changes represent an increased need for assistance with daily activities.
Time Frame: Baseline to Weeks 12, 24, 36, 48, 60, 72, 84
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | SC TCZ Q2W | SC TCZ QW
Number analyzed (Participants) | 44 | 173
units on a scale
  Week 12 (n=44,172) | -0.02 (0.254) | -0.10 (0.339)
  Week 24 (n=43,167) | -0.01 (0.272) | -0.11 (0.372)
  Week 36 (n=39,159) | -0.08 (0.276) | -0.09 (0.394)
  Week 48 (n=18,141) | -0.01 (0.237) | -0.14 (0.390)
  Week 60 (n=2,92) | 0.56 (0.795) | -0.08 (0.394)
  Week 72 (n=1,52) | 0.88 (NA) — Standard deviation could not be calculated because the analysis only included 1 participant. | -0.06 (0.420)
  Week 84 (n=0,11) | NA (NA) — No participants provided evaluable data for the analysis | -0.07 (0.397)

36. Secondary Outcome: Percentage of Participants With HAQ-DI Score <0.5
Description: The Stanford HAQ-DI was calculated as the average of 20 questions, each scored from 0 (no difficulty) to 3 (unable to do). The questionnaire included 8 component sets: dressing/grooming, arising, eating, walking, hygiene, reach, grip, and common activities. Overall scores may range from 0 to 3, with higher scores representing increased disability. The percentage of participants achieving a score <0.5 was calculated at each visit.
Time Frame: Baseline and Weeks 12, 24, 36, 48, 60, 72, 84
Population: ITT Population; only those participants who provided evaluable data (n) were included in the analysis.
Measure: Number; unit: percentage of participants
Arm/Group | SC TCZ Q2W | SC TCZ QW
Number analyzed (Participants) | 44 | 173
percentage of participants
  Baseline (n=44,173) | 31.8 | 17.9
  Week 12 (n=44,172) | 27.3 | 20.9
  Week 24 (n=43,167) | 32.6 | 23.4
  Week 36 (n=39,159) | 38.5 | 24.5
  Week 48 (n=18,141) | 27.8 | 24.8
  Week 60 (n=2,92) | 0.0 | 29.3
  Week 72 (n=1,52) | 0.0 | 34.6
  Week 84 (n=0,11) | NA — No participants provided evaluable data for the analysis | 9.1

37. Secondary Outcome: Number of Participants With Low Disease Activity According to DAS28, SDAI, and CDAI Criteria
Description: Low disease activity was defined as DAS28 ≤3.2, SDAI ≤11, or CDAI ≤10. For each formula, the SJC and TJC values were based upon 28 joints, and VAS was transformed from a 100-mm scale to a 10-point score. The DAS28 was calculated as (0.56 × square root of TJC) + (0.28 × square root of SJC) + (0.7 × ln ESR) + (0.014 × VAS), with potential scores from 0 to 10. The SDAI was calculated as SJC + TJC + VAS (participant) + VAS (physician) + hsCRP, with potential scores from 0 to infinity. However, based upon normal hsCRP level within 1 mg/dL, scores would be expected to fall within ≤77 points. The CDAI was calculated as SJC + TJC + VAS (participant) + VAS (physician), with potential scores from 0 to 76. For all instruments, higher scores indicate increased disease activity. The number of participants who met criteria for low disease activity was reported at each visit.
Time Frame: Baseline and Weeks 12, 24, 36, 48, 60, 72, 84
Population: ITT Population; only those participants who provided evaluable data (n) were included in the analysis.
Measure: Number; unit: participants
Arm/Group | SC TCZ Q2W | SC TCZ QW
Number analyzed (Participants) | 44 | 173
participants
  Baseline, DAS28 (n=44,172) | 11 | 46
  Baseline, SDAI (n=44,170) | 14 | 43
  Baseline, CDAI (n=44,173) | 13 | 41
  Week 12, DAS28 (n=44,172) | 21 | 81
  Week 12, SDAI (n=44,172) | 22 | 65
  Week 12, CDAI (n=44,172) | 20 | 63
  Week 24, DAS28 (n=43,168) | 23 | 82
  Week 24, SDAI (n=41,166) | 19 | 67
  Week 24, CDAI (n=42,166) | 20 | 60
  Week 36, DAS28 (n=39,159) | 21 | 75
  Week 36, SDAI (n=39,159) | 20 | 61
  Week 36, CDAI (n=39,159) | 21 | 60
  Week 48, DAS28 (n=18,141) | 10 | 69
  Week 48, SDAI (n=18,140) | 8 | 63
  Week 48, CDAI (n=18,140) | 7 | 59
  Week 60, DAS28 (n=2,92) | 0 | 52
  Week 60, SDAI (n=2,92) | 0 | 40
  Week 60, CDAI (n=2,92) | 0 | 37
  Week 72, DAS28 (n=1,52) | 0 | 28
  Week 72, SDAI (n=1,52) | 0 | 26
  Week 72, CDAI (n=1,52) | 0 | 25
  Week 84, DAS28 (n=0,11) | NA — No participants provided evaluable data for the analysis | 6
  Week 84, SDAI (n=0,11) | NA — No participants provided evaluable data for the analysis | 4
  Week 84, CDAI (n=0,11) | NA — No participants provided evaluable data for the analysis | 4

38. Secondary Outcome: Percentage of Participants With Low Disease Activity According to DAS28, SDAI, and CDAI Criteria
Description: Low disease activity was defined as DAS28 ≤3.2, SDAI ≤11, or CDAI ≤10. For each formula, the SJC and TJC values were based upon 28 joints, and VAS was transformed from a 100-mm scale to a 10-point score. The DAS28 was calculated as (0.56 × square root of TJC) + (0.28 × square root of SJC) + (0.7 × ln ESR) + (0.014 × VAS), with potential scores from 0 to 10. The SDAI was calculated as SJC + TJC + VAS (participant) + VAS (physician) + hsCRP, with potential scores from 0 to infinity. However, based upon normal hsCRP level within 1 mg/dL, scores would be expected to fall within ≤77 points. The CDAI was calculated as SJC + TJC + VAS (participant) + VAS (physician), with potential scores from 0 to 76. For all instruments, higher scores indicate increased disease activity. The percentage of participants who met criteria for low disease activity was calculated at each visit.
Time Frame: Baseline and Weeks 12, 24, 36, 48, 60, 72, 84
Population: ITT Population; only those participants who provided evaluable data (n) were included in the analysis.
Measure: Number; unit: percentage of participants
Arm/Group | SC TCZ Q2W | SC TCZ QW
Number analyzed (Participants) | 44 | 173
percentage of participants
  Baseline, DAS28 (n=44,172) | 25.0 | 26.7
  Baseline, SDAI (n=44,170) | 31.8 | 25.3
  Baseline, CDAI (n=44,173) | 29.5 | 23.7
  Week 12, DAS28 (n=44,172) | 47.7 | 47.1
  Week 12, SDAI (n=44,172) | 50.0 | 37.8
  Week 12, CDAI (n=44,172) | 45.5 | 36.6
  Week 24, DAS28 (n=43,168) | 53.5 | 48.8
  Week 24, SDAI (n=41,166) | 46.3 | 40.4
  Week 24, CDAI (n=42,166) | 47.6 | 36.1
  Week 36, DAS28 (n=39,159) | 53.8 | 47.2
  Week 36, SDAI (n=39,159) | 51.3 | 38.4
  Week 36, CDAI (n=39,159) | 53.8 | 37.7
  Week 48, DAS28 (n=18,141) | 55.6 | 48.9
  Week 48, SDAI (n=18,140) | 44.4 | 45.0
  Week 48, CDAI (n=18,140) | 38.9 | 42.1
  Week 60, DAS28 (n=2,92) | 0.0 | 56.5
  Week 60, SDAI (n=2,92) | 0.0 | 43.5
  Week 60, CDAI (n=2,92) | 0.0 | 40.2
  Week 72, DAS28 (n=1,52) | 0.0 | 53.8
  Week 72, SDAI (n=1,52) | 0.0 | 50.0
  Week 72, CDAI (n=1,52) | 0.0 | 48.1
  Week 84, DAS28 (n=0,11) | NA — No participants provided evaluable data for the analysis | 54.5
  Week 84, SDAI (n=0,11) | NA — No participants provided evaluable data for the analysis | 36.4
  Week 84, CDAI (n=0,11) | NA — No participants provided evaluable data for the analysis | 36.4

39. Secondary Outcome: Number of Participants With Remission According to DAS28, SDAI, and Boolean Criteria
Description: Remission was defined as DAS28 <2.6, SDAI ≤3.3, or meeting all Boolean criteria (28-count SJC and TJC ≤1, VAS ≤10 mm, and hsCRP ≤1 mg/dL). For DAS28 and SDAI formulas, the SJC and TJC values were based upon 28 joints, and VAS was transformed from a 100-mm scale to a 10-point score. The DAS28 was calculated as (0.56 × square root of TJC) + (0.28 × square root of SJC) + (0.7 × ln ESR) + (0.014 × VAS), with potential scores from 0 to 10. The SDAI was calculated as SJC + TJC + VAS (participant) + VAS (physician) + hsCRP, with potential scores from 0 to infinity. However, based upon normal hsCRP level within 1 mg/dL, scores would be expected to fall within ≤77 points. For these instruments, higher scores indicate increased disease activity. The number of participants who met criteria for remission was reported at each visit.
Time Frame: Baseline and Weeks 12, 24, 36, 48, 60, 72, 84
Population: as for outcome 7
Measure: Number; unit: participants
Arm/Group | SC TCZ Q2W | SC TCZ QW
Number analyzed (Participants) | 44 | 173
participants
  Baseline, DAS28 (n=44,172) | 6 | 33
  Baseline, SDAI (n=44,170) | 2 | 15
  Baseline, Boolean (n=44,172) | 1 | 14
  Week 12, DAS28 (n=44,172) | 14 | 61
  Week 12, SDAI (n=44,172) | 7 | 20
  Week 12, Boolean (n=44,172) | 4 | 15
  Week 24, DAS28 (n=43,168) | 18 | 61
  Week 24, SDAI (n=41,166) | 8 | 23
  Week 24, Boolean (n=43,170) | 5 | 16
  Week 36, DAS28 (n=39,159) | 15 | 57
  Week 36, SDAI (n=39,159) | 7 | 21
  Week 36, Boolean (n=39,161) | 3 | 17
  Week 48, DAS28 (n=18,141) | 9 | 51
  Week 48, SDAI (n=18,140) | 1 | 15
  Week 48, Boolean (n=18,143) | 1 | 14
  Week 60, DAS28 (n=2,92) | 0 | 39
  Week 60, SDAI (n=2,92) | 0 | 17
  Week 60, Boolean (n=2,93) | 0 | 14
  Week 72, DAS28 (n=1,52) | 0 | 22
  Week 72, SDAI (n=1,52) | 0 | 11
  Week 72, Boolean (n=1,54) | 0 | 10
  Week 84, DAS28 (n=0,11) | NA — No participants provided evaluable data for the analysis | 6
  Week 84, SDAI (n=0,11) | NA — No participants provided evaluable data for the analysis | 2
  Week 84, Boolean (n=0,11) | NA — No participants provided evaluable data for the analysis | 2

40. Secondary Outcome: Percentage of Participants With Remission According to DAS28, SDAI, and Boolean Criteria
Description: Remission was defined as DAS28 <2.6, SDAI ≤3.3, or meeting all Boolean criteria (28-count SJC and TJC ≤1, VAS ≤10 mm, and hsCRP ≤1 mg/dL). For DAS28 and SDAI formulas, the SJC and TJC values were based upon 28 joints, and VAS was transformed from a 100-mm scale to a 10-point score. The DAS28 was calculated as (0.56 × square root of TJC) + (0.28 × square root of SJC) + (0.7 × ln ESR) + (0.014 × VAS), with potential scores from 0 to 10. The SDAI was calculated as SJC + TJC + VAS (participant) + VAS (physician) + hsCRP, with potential scores from 0 to infinity. However, based upon normal hsCRP level within 1 mg/dL, scores would be expected to fall within ≤77 points. For these instruments, higher scores indicate increased disease activity. The percentage of participants who met criteria for remission was calculated at each visit.
Time Frame: Baseline and Weeks 12, 24, 36, 48, 60, 72, 84
Population: as for outcome 7
Measure: Number; unit: percentage of participants
Arm/Group | SC TCZ Q2W | SC TCZ QW
Number analyzed (Participants) | 44 | 173
percentage of participants
  Baseline, DAS28 (n=44,172) | 13.6 | 19.2
  Baseline, SDAI (n=44,170) | 4.5 | 8.8
  Baseline, Boolean (n=44,172) | 2.3 | 8.1
  Week 12, DAS28 (n=44,172) | 31.8 | 35.5
  Week 12, SDAI (n=44,172) | 15.9 | 11.6
  Week 12, Boolean (n=44,172) | 9.1 | 8.7
  Week 24, DAS28 (n=43,168) | 41.9 | 36.3
  Week 24, SDAI (n=41,166) | 19.5 | 13.9
  Week 24, Boolean (n=43,170) | 11.6 | 9.4
  Week 36, DAS28 (n=39,159) | 38.5 | 35.8
  Week 36, SDAI (n=39,159) | 17.9 | 13.2
  Week 36, Boolean (n=39,161) | 7.7 | 10.6
  Week 48, DAS28 (n=18,141) | 50.0 | 36.2
  Week 48, SDAI (n=18,140) | 5.6 | 10.7
  Week 48, Boolean (n=18,143) | 5.6 | 9.8
  Week 60, DAS28 (n=2,92) | 0.0 | 42.4
  Week 60, SDAI (n=2,92) | 0.0 | 18.5
  Week 60, Boolean (n=2,93) | 0.0 | 15.1
  Week 72, DAS28 (n=1,52) | 0.0 | 42.3
  Week 72, SDAI (n=1,52) | 0.0 | 21.2
  Week 72, Boolean (n=1,54) | 0.0 | 18.5
  Week 84, DAS28 (n=0,11) | NA — No participants provided evaluable data for the analysis | 54.5
  Week 84, SDAI (n=0,11) | NA — No participants provided evaluable data for the analysis | 18.2
  Week 84, Boolean (n=0,11) | NA — No participants provided evaluable data for the analysis | 18.2

ADVERSE EVENTS:
Time Frame: From Baseline to 8 weeks after last dose; assessed continuously during treatment (up to 96 weeks) and up to 8 weeks after last dose (up to 2 years overall)
Description: Safety Population.
Arm/Group | SC TCZ Q2W | SC TCZ QW
Serious Adverse Events (participants affected / at risk) | 4/44 | 19/173
Other Adverse Events (participants affected / at risk) | 22/44 | 102/173
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | SC TCZ Q2W (N=44) | SC TCZ QW (N=173)
Cellulitis (Infections and infestations) | 0 | 2
Staphylococcal bacteraemia (Infections and infestations) | 0 | 2
Arthritis bacterial (Infections and infestations) | 0 | 1
Bronchopneumonia (Infections and infestations) | 0 | 1
Endocarditis (Infections and infestations) | 0 | 1
Endophthalmitis (Infections and infestations) | 1 | 0
Pyelonephritis (Infections and infestations) | 1 | 0
Syncope (Nervous system disorders) | 1 | 1
Transient ischaemic attack (Nervous system disorders) | 0 | 2
Cerebrovascular accident (Nervous system disorders) | 0 | 1
Abdominal compartment syndrome (Gastrointestinal disorders) | 1 | 0
Diverticular perforation (Gastrointestinal disorders) | 0 | 1
Gastric ulcer perforation (Gastrointestinal disorders) | 0 | 1
Pancreatitis (Gastrointestinal disorders) | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Chest pain (General disorders) | 0 | 1
Device malfunction (General disorders) | 0 | 1
Joint dislocation (Injury, poisoning and procedural complications) | 0 | 1
Post procedural complication (Injury, poisoning and procedural complications) | 0 | 1
Deep vein thrombosis (Vascular disorders) | 1 | 0
Hypertension (Vascular disorders) | 0 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 1
Endometrial stromal sarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Mental status change (Psychiatric disorders) | 0 | 1
Haematuria (Renal and urinary disorders) | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Drug eruption (Skin and subcutaneous tissue disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | SC TCZ Q2W (N=44) | SC TCZ QW (N=173)
Upper respiratory tract infection (Infections and infestations) | 8 | 35
Sinusitis (Infections and infestations) | 2 | 22
Nasopharyngitis (Infections and infestations) | 2 | 20
Urinary tract infection (Infections and infestations) | 2 | 15
Bronchitis (Infections and infestations) | 1 | 11
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 12
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 9
Fall (Injury, poisoning and procedural complications) | 3 | 6
Contusion (Injury, poisoning and procedural complications) | 3 | 5
Alanine aminotransferase increased (Investigations) | 0 | 12
Diarrhoea (Gastrointestinal disorders) | 3 | 8
Rash (Skin and subcutaneous tissue disorders) | 3 | 6
Hypertension (Vascular disorders) | 0 | 9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.